CLINICAL TRIAL: NCT00324233
Title: Evaluation of Residual Urine After Intermittent Catheterisation - Comparison of 2 Hydrophilic Coated, Intermittent Catheters
Brief Title: Evaluation of Residual Urine After Intermittent Catheterisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DK052CC
Record Dates: First submitted 2006-05-09; First posted 2006-05-10 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2013-01-01 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Residual urine; Hematuria; Ultra sound
MeSH Terms: conditions — Hematuria

ARMS (2):
- SC (Active Comparator): Speedicath (SC) catheter is a catheter for intermittent catherisation
  Interventions: Device: Intermittent catheter
- SCCM (Experimental): SpeediCath Compact Male (SCCM) is a compact catheter for intermittent catherisation to be used by males
  Interventions: Device: Compact intermittent catheter

INTERVENTIONS:
Device: Intermittent catheter — SpeediCath catherter (SC) for intermittent catherisation
  Arms: SC
Device: Compact intermittent catheter — SpeediCath Compact Male catheter (SCCM) is a compact intermittent catheter for males
  Arms: SCCM

SUMMARY:
Intermittent catheterization is a well-known method used for emptying the bladder. The objective of this study is to compare the residual urine after intermittent catheterisation with 2 different, hydrophilic coated, intermittent catheters. The study is a randomized, single blinded, crossover study including 24 healthy males.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18 years and above
* A negative urine dip-stick
* Have signed informed written consent to participate

Exclusion Criteria:

* The test participant has previous or current congenital deformity, diseases or operation in the lower urinary tract

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Bagi, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, København Ø, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- SC Then SCCM: SpeediCath (SC)catheter in first period then SpeediCath Compact Male (SCCM)catheter in second period
- SCCM Then SC: SpeediCath Compact Male (SCCM)catheter in the first period then SpeediCath(SC)catheter in second period
Period: First Period
Arm/Group | SC Then SCCM | SCCM Then SC
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — unable to insert catheter | 1 | 0
Period: Second Period
Arm/Group | SC Then SCCM | SCCM Then SC
Started | 17 | 18
Completed | 12 | 11
Not Completed | 5 | 7
Not completed — unable to insert catheter | 1 | 1
Not completed — Protocol Violation | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SC Then SCCM | SCCM Then SC | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.6 (3.0) | 23.9 (2.9) | 23.7 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  Denmark | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Residual Urine Measured by Ultra Sound
Time Frame: 2
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | SpeediCath | SpediCath Compact Male
Number analyzed (Participants) | 36 | 33
ml | 11 (30) | 6 (23)
Statistical Analysis 1: Comparison: SpeediCath vs SpediCath Compact Male; Test type: Superiority or Other; p = 0.56, equivalence testing

2. Secondary Outcome: Subjectively Measured Handling
Reporting Status: Not Posted

3. Secondary Outcome: Subjectively Measured Insertion of the Catheter
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | SC Then SCCM | SCCM Then SC
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less